CLINICAL TRIAL: NCT03516617
Title: Randomized Phase 2 Study Comparing Acalabrutinib to Acalabrutinib and Obinutuzumab in the Treatment of Patients With Early-Stage Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma (CLL/SLL) Who Are at High Risk of Disease Progression
Brief Title: Acalabrutinib With or Without Obinutuzumab in Treating Patients With Early-Stage Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC168E; NCI-2018-00591 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17-008161 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2018-04-23; First posted 2018-05-04 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — acalabrutinib; obinutuzumab; Watchful Waiting; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (acalabrutinib) (Experimental): Patients receive acalabrutinib PO BID on days 1-28. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive acalabrutinib PO BID on days 1-84. Treatment repeats every 84 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue treatment with acalabrutinib If MRD negative CR/CRi is not achieved after 12 cycles.
  Interventions: Drug: Acalabrutinib; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment
- Arm B (acalabrutinib, obinutuzumab) (Experimental): Patients receive acalabrutinib PO BID on days 1-28 and obinutuzumab IV on days 1, 2, 8, and 15 of cycle 1 and days 1 of subsequent cycles. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive acalabrutinib PO BID on days 1-84. Treatment repeats every 84 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue treatment with acalabrutinib If MRD negative CR/CRi is not achieved after 12 cycles.
  Interventions: Drug: Acalabrutinib; Other: Laboratory Biomarker Analysis; Biological: Obinutuzumab; Other: Quality-of-Life Assessment
- Arm C (observation) (Active Comparator): Patients will be observed every 6 months for up to 2 years.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Patient Observation; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Acalabrutinib — Given PO
  Other Names: ACP-196; Bruton Tyrosine Kinase Inhibitor ACP-196
  Arms: Arm A (acalabrutinib); Arm B (acalabrutinib, obinutuzumab)
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Obinutuzumab — Given IV
  Other Names: Anti-CD20 Monoclonal Antibody R7159; GA-101; GA101; Gazyva; huMAB(CD20); R7159; RO 5072759; RO-5072759; RO5072759
  Arms: Arm B (acalabrutinib, obinutuzumab)
Other: Patient Observation — Undergo observation
  Other Names: Active Surveillance; deferred therapy; expectant management; Observation; Watchful Waiting
  Arms: Arm C (observation)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This phase II trials studies how well acalabrutinib with or without obinutuzumab works in treating patients with early-stage chronic lymphocytic leukemia or small lymphocytic lymphoma. Acalabrutinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as obinutuzumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. It is not yet known whether giving acalabrutinib with or without obinutuzumab will work better in treating patients with early-stage chronic lymphocytic leukemia or small lymphocytic lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the bone marrow minimal residual disease (MRD)-negative complete response (CR) rate of acalabrutinib alone and acalabrutinib/obinutuzumab in early stage asymptomatic chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL) patients who are high and very high risk by CLL-International Prognostic Index (IPI). (Arms A and B) II. To evaluate time to first therapy (TFT) in early stage asymptomatic CLL/SLL patients with low and intermediate-risk by CLL-IPI. (Arm C)

SECONDARY OBJECTIVES:

I. To compare the safety of acalabrutinib alone and acalabrutinib/obinutuzumab in early stage asymptomatic CLL/SLL patients who are high and very high risk by CLL-IPI.

II. To compare the overall response rate (ORR), progression-free survival (PFS), time to next therapy (TNT) and overall survival (OS) of acalabrutinib alone and acalabrutinib/obinutuzumab in early stage asymptomatic CLL/SLL patients who are at high and very high risk by CLL-IPI.

III. To determine the progression-free survival (PFS) and overall survival (OS) in early stage asymptomatic CLL/SLL patients with low and intermediate risk by CLL-IPI.

EXPLORATORY OBJECTIVE:

I. To evaluate the quality of life using Functional Assessment of Cancer Therapy-General (FACT-G) quality of life (QOL) survey.

CORRELATIVE RESEARCH:

I. To compare the peripheral blood immune profile using 8-color flow cytometry, to assess changes in T-cells, natural killer (NK)-cells, and NK-T cells at baseline and during active treatment among patients receiving either acalabrutinib alone or acalabrutinib and obinutuzumab.

II. To determine changes in the peripheral blood immune profile using 8-color flow cytometry to assess changes in T-cells, NK-cells, and NK-T cells at baseline and during event monitoring in patients with low and intermediate risk by CLL-IPI.

III. Signal pathway studies-BTK, ERK, PLC gamma and S6 protein levels and phosphorylation status will be assessed by Western blot methodology using specific antibodies to pull down specific proteins from cell lysates.

IV. To confirm if in vitro cell killing is via apoptosis we will also assess PARP and caspase 3 cleavage.

V. Apoptotic protein studies-MCL-1, XIAP levels will be determined by Western blot methodology using specific antibodies to pull down these specific proteins from cell lysates.

VI. Bone marrow aspirates will be studied for hematopoietic function in two ways:

VIa. Estimation of colony forming capacity by purified hematopoietic stem cells (HSCs).

VIb. Evaluation of the levels of HSCs and their differentiated progeny (i.e. MPP, CMP, CLP).

VII. Paired bone marrow and blood samples will be evaluated for the levels of innate effector cells.

VIII. Perform targeted sequencing of 59 genes mainly grouped in 8 biological pathways: NOTCH1, B-cell signaling, deoxyribonucleic acid (DNA) damage response, chromatin modifiers, ribonucleic acid (RNA) metabolism, NF-kappaB pathway, cell cycle and apoptosis.

IX. Screen 2 genes previously associated with resistance to BTK inhibitors (BTK and PLCG2).

OUTLINE: Patients with high or very high risk CLL-IPI are randomized to Arm A or Arm B. Patients with intermediate or low risk are assigned to Arm C.

ARM A: Patients receive acalabrutinib orally (PO) twice daily (BID) on days 1-28. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive acalabrutinib PO BID on days 1-84. Treatment repeats every 84 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue treatment with acalabrutinib If MRD negative CR/CR with incomplete marrow recovery (CRi) is not achieved after 12 cycles.

ARM B: Patients receive acalabrutinib orally (PO) twice daily (BID) on days 1-28 and obinutuzumab intravenously (IV) on days 1, 2, 8, and 15 of cycle 1 and days 1 of subsequent cycles. Treatment repeats every 28 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then receive acalabrutinib PO BID on days 1-84. Treatment repeats every 84 days for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients may continue treatment with acalabrutinib If MRD negative CR/CRi is not achieved after 12 cycles.

ARM C: Patients will be observed every 6 months for up to 2 years.

After completion of study treatment, patients are followed up every 6 months for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Diagnosis of:

  * Biopsy-proven small lymphocytic lymphoma (SLL) , or
  * Diagnosis of chronic lymphocytic leukemia (CLL) with a clonal B-cell population in the peripheral blood with immunophenotyping consistent with CLL as follows:

    * The population of lymphocytes share both B-cell antigens (CD19, CD20 [typically dim expression], or CD23) as well as CD5 in the absence of other pan-T-cell markers (CD3, CD2, etc.)
    * Clonality as evidenced by kappa or lambda light chain expression (typically dim immunoglobulin expression) or other genetic method (e.g. IGHV analysis)
    * Before diagnosing CLL or SLL, mantle cell lymphoma must be excluded by demonstrating a negative fluorescence in situ hybridization (FISH) analysis for t(11;14)(IgH/CCND1)
* Patients must be previously untreated

  * Note: Prior chemotherapy or monoclonal antibody based therapy for treatment of CLL or SLL will be considered prior therapy; nutraceutical treatments with no established benefit in CLL (such as epigallocatechin gallate or EGCG, found in green tea or other herbal treatments or supplemental vitamins) will not be considered "prior treatment"; prior corticosteroid therapy for an indication other than CLL/SLL will not be considered "prior treatment"
* All patients will undergo testing for prognostic factors according to the CLL-IPI (testing obtained =< 730 days prior to registration)

  * Note: If the results for any of the prognostic factors included in the CLL-IPI are unknown including IGVH mutation status results not being available due to a failed laboratory assay, the patient is not eligible
  * Note: When determining CLL-IPI, use most recent test results, if more than one result is available
  * Note: Patients with CLL-IPI risk category of high risk or very high risk (total score of 4-10) will be randomized to Arms A or B
  * Note: Patients with CLL-IPI risk category of low risk or intermediate risk (total score of 0-3) will be registered to Arm C
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2
* Provide written informed consent
* Willing to provide blood and saliva samples for correlative research purposes
* Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* For high risk and very high risk CLL-IPI (Arms A and B) only: Absolute neutrophil count (ANC) >= 1500/mm^3 (obtained =< 30 days prior to randomization)
* For high risk and very high risk CLL-IPI (Arms A and B) only: Platelet count >= 100,000/mm^3 (obtained =< 30 days prior to randomization)
* For high risk and very high risk CLL-IPI (Arms A and B) only: Hemoglobin >= 11.0 g/dL (obtained =< 30 days prior to randomization)
* For high risk and very high risk CLL-IPI (Arms A and B) only: Aspartate aminotransferase (aspartate transaminase [AST]) =< 3 x upper limit of normal (ULN) (obtained =< 30 days prior to randomization)
* For high risk and very high risk CLL-IPI (Arms A and B) only: Creatinine =< 1.5 X ULN (obtained =< 30 days prior to randomization)
* For high risk and very high risk CLL-IPI (Arms A and B) only: Total bilirubin =< 1.5 x upper limit of normal (ULN) (or total bilirubin =< 3.0 x ULN with direct bilirubin =< 1.5 x ULN in patients with well-documented Gilbert's syndrome (obtained =< 30 days prior to randomization)
* For high risk and very high risk CLL-IPI (Arms A and B) only: Prothrombin time (PT), international normalized ratio (INR), and partial thromboplastin time (PTT) =< 1.5 X ULN OR if patient is receiving anticoagulant therapy and PT or PTT is within therapeutic range of intended use of coagulants (obtained =< 30 days prior to randomization)
* Negative serum pregnancy test done =< 7 days prior to registration, for persons of childbearing potential only
* Will provide bone marrow aspirate sample for correlative research purposes

Exclusion Criteria:

* Date of CLL/SLL diagnosis >= 24 months prior to registration
* Prior exposure to ibrutinib or to a BCR inhibitor (e.g. Btk or PI3 kinase or Syk inhibitors) or a BCL-2 inhibitor (e.g. venetoclax)
* Known central nervous system (CNS) lymphoma or leukemia
* Patients with any of the following indications for chemotherapy:

  * Evidence of progressive marrow failure as manifested by the development of or worsening anemia (=< 11 g/dL) and/or thrombocytopenia (=< 100 x 10^9/L) not due to autoimmune disease
  * Symptomatic or progressive lymphadenopathy, splenomegaly or hepatomegaly
  * One or more of the following disease-related symptoms:

    * Weight loss >= 10% within the previous 6 months
    * Extreme fatigue attributed to CLL
    * Fevers >= 100.4 degrees Fahrenheit (F) for 2 weeks without evidence of infection
    * Drenching night sweats without evidence of infection
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy; NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy =< 2 years prior to registration; EXCEPTIONS: Non-melanotic skin cancer, carcinoma-in-situ of the cervix, or early stage prostate cancer
* History of myocardial infarction =< 6 months prior to registration, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* For high risk and very high risk CLL-IPI (Arms A and B) only:

  * Any of the following:

    * Pregnant persons
    * Nursing persons
    * Persons of childbearing potential who are unwilling to employ highly effective contraception
  * Serologic status reflecting active hepatitis B or C infection

    * NOTE: Subjects with hepatitis B core antibody positive who are surface antigen negative or who are hepatitis C antibody positive will need to have a negative polymerase chain reaction (PCR) result before randomization; those who are hepatitis B surface antigen positive or hepatitis B PCR positive and those who are hepatitis C PCR positive will be excluded
  * History of stroke or intracranial hemorrhage within 6 months before randomization
  * History of bleeding diathesis (e.g. hemophilia, von Willebrand disease)
  * Requires or receiving anticoagulation with warfarin or equivalent vitamin K antagonists (e.g. phenprocoumon) within 7 days of first dose of study drug and while on study
  * Requires treatment with a strong CYP3A inducer
  * Presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months before screening
  * History of confirmed progressive multifocal leukoencephalopathy (PML)
  * Received a vaccination with a live vaccine =< 28 days prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-09-10 (Actual); Primary Completion 2027-03-15 (Estimated); Study Completion 2030-10-16 (Estimated)

PRIMARY OUTCOMES:
Rate of minimal residual disease (MRD)-negative complete response (Arm A and Arm B) | After 12 cycles (cycle 1-6 = 28 days, cycles 7 and beyond = 84 days)
  Defined as an objective status of complete response (CR) or CR with incomplete marrow recovery (CRi) along with MRD negativity in the bone marrow by flow cytometry. Will be compared between the two arms. The proportion of successes will be estimated in each arm by the number of successes divided by the total number of evaluable patients. Ninety-five percent confidence intervals for the true success proportion will be calculated in each arm based on the normal approximation. Comparison of MRD-negative complete response rates between the two treatment groups will be performed using a one-sided z-test (based on normal approximation with pooled variance of standardized test statistics) at significance level 0.10.
Time to first therapy (TFT) in patients (Arm C) | After 12 cycles (one cycle = 6 months)
  Defined as the time from the date of registration to the date of initiation of treatment for CLL.

SECONDARY OUTCOMES:
Overall response rate (Arms A and B) | Up to 10 years
  Will be assessed in each arm by the number of patients who achieve complete remission (CR), complete remission with incomplete count recovery (CRi), clinical complete response (CCR), nodular partial response (nPR), or partial response (PR) at any time during treatment.
Progression-free survival (Arms A and B) | From randomization up to 10 years
  Defined as the time from randomization to the earliest date of documentation of disease progression or death due to any cause.
Time to next therapy (Arms A and B) | From the date of randomization up to 10 years
  Defined as the time from the date of randomization to the date of initiation of subsequent treatment for CLL.
Overall survival (Arms A and B) | From randomization up to 10 years
  Defined as the time from randomization until death due to any cause.
Progression-free survival (Arm C) | From randomization up to 10 years
  Defined as the time from randomization to the earliest date of documentation of disease progression or death due to any cause.
Overall survival (Arm C) | From randomization up to 10 years
  Defined as the time from randomization until death due to any cause.
Incidence of adverse events rates (Arms A and B) | Up to 10 years
  Will be assessed according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed for each arm to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.

OTHER OUTCOMES:
Quality of life | Up to 10 years
  Will be assessed using the Functional Assessment of Cancer Therapy-General (FACT-G), a 27-item questionnaire that measures Health-related quality of life (HRQoL) in cancer patients. Responses to each question are scored on a 5-point Likert scale ranging from 0 (Not at all) to 4 (Very much). Possible total scores range from 0-108, with higher scores indicating a better outcome/better quality QOL.
T-cells, natural killer (NK)-cells, and NK-T cells | Baseline
  Will be assessed in peripheral blood immune profile using 8-color flow cytometry. Values over time will be summarized graphically and descriptively. Paired sample approaches (Wilcoxon signed rank test) for these types of quantitative measures will be used to assess differences over time. Differences between treatments (Arms A and B only) will be assessed.
Bone marrow hematopoiesis (Arms A and B) | Up to 10 years
  will be evaluated by estimation of colony forming capacity by purified hematopoietic stem cells (HSCs) and their differentiated progeny (i.e. multipotent progenitor, common myeloid progenitor, common lymphoid progenitor) as continuous measures. Degree of cytopenia in the peripheral blood will be evaluated on a continuous scale for each blood cell component (hemoglobin, platelets, etc.). In each arm, correlation between each blood cell component and its corresponding pre-cursor will be evaluated using Spearman's rank correlation coefficients.
Percent killing of chronic lymphocytic leukemia (CLL) B-cells (Arms A and B) | After 12 courses
  Will be measured as a continuous measure. In each arm, the relationship between percent killing and response (responder versus [vs.] non-responder) after 12 cycles of treatment will be evaluating using Wilcoxon's rank sum test.
Somatic genetic mutations (Arms A and B) | After 12 courses
  Will be evaluated as present vs. absent for each gene. In each arm, the relationship between each mutation and response (responder vs. non-responder) after 12 cycles of treatment will be evaluated using Fisher's exact test.

CONTACTS AND LOCATIONS:
Overall Officials: Sameer A. Parikh, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials